CLINICAL TRIAL: NCT04763356
Title: Remote Monitoring and Management of Chemotherapy Induced Peripheral Neuropathy
Acronym: REMOTE-CIPN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Virginia Commonwealth University (Other); University of Utah (Other)
Responsible Party: Principal Investigator, Noah Kolb, Principal Investigator, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REMOTECIPN1
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-03

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy

STUDY DESIGN:
Intervention Model Description: This is a single blinded (outcome assessor) randomized controlled trial with 2 arms.
Who Masked: Outcomes Assessor
Masking Description: The assessor grading the only reported outcome measure (mTCNS) will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (UC) (No Intervention): The UC group (control) models the current standard of care model. The NTSS-6 will be completed daily by participants using the SCH system. The results will not be reported to their oncology team. Participants will be counseled at study entry to contact their treating care team to manage CIPN symptoms. They will also receive a reminder to do so at the end of each reporting session. UC participants will attend all regular visits with these providers and can receive any type of treatment for their CIPN symptoms. There are no limitations on the therapies that can be prescribed, or the means by which the clinical team communicates with the participant. Treating physicians will be provided with links to the current ASCP and NCCN guidelines but will not be provided with the algorithm as this group is meant to reflect current standard medical practice.
- SCH with NP follow-up (SCH-NP) (Experimental): Participants will report daily symptom as above. The SCH system will notify the study NP for any of the following symptoms measured by the NTSS6: aching, allodynia, burning, lancinating, numbness, and prickling that are concerning. Participants will receive a NP call back either the same day or the next day, depending on the time they reported their symptoms. The NP will follow a standardized script to elicit details about the CIPN symptoms and recommend and prescribe CIPN treatment per the treatment algorithm.
  Interventions: Other: Symptom Care at Home with NP follow up

INTERVENTIONS:
Other: Symptom Care at Home with NP follow up — In the SCH-NP group all participants will report their CIPN related symptoms daily via the app, website or phone tree. Any concerning symptoms will trigger a call back from a nurse practitioner who will use a consensus and evidence based algorithm to prescribe therapies for the CIPN symptoms.
  Arms: SCH with NP follow-up (SCH-NP)

SUMMARY:
This is a prospective randomized trial designed to investigate a new care model for patients who suffer from nerve damage from chemotherapy called chemotherapy induced peripheral neuropathy (CIPN). All participants in the study will report their CIPN symptoms daily using a website, app or phone for 12 weeks. In one group the data will be collected and participants will be encouraged to reach out to their treating doctors for uncontrolled symptoms. These participants' doctors can prescribe any treatment they feel is appropriate. In the second group, if the symptoms meet the criteria for eligibility they will receive a phone call from a nurse practitioner either the same day or next day, depending on the time symptoms were logged. That nurse practitioner will determine the correct CIPN treatment using an algorithm and prescribe it. The study will track the severity of symptoms over time as well as looking at the impact on treatments for CIPN (medications and referrals).

DETAILED DESCRIPTION:
This is a prospective single blinded (outcome assessor) randomized controlled trial of a CIPN care model that pairs a personalized suite of remote symptom monitoring technologies with triggered real time responses from a nurse practitioner (NP) equipped to enact algorithmic guideline based CIPN treatment in response to poorly controlled symptoms. The study will enroll adult cancer patients who have, within the last 540 days, completed a course of a taxane, platinum, or vinca alkaloid-based agent, bortezomib, thalidomide, lenalidomide, ixazomib or brentuximab vedotin, or have been receiving ongoing maintenance therapy with bortezomib, thalidomide, lenalidomide or ixazomib for >90 days, and have been diagnosed with CIPN. Participants will log neuropathy symptoms daily for a one week run-in period using a remote symptom monitoring technology described below. Participants who meet the criteria to proceed in the study will be randomized in a 1:1 ratio to Usual Care (UC) or Symptom Care at Home with Nurse Practitioner follow up (SCH-NP). Those not meeting eligibility criteria will be excluded but can be rescreened 6 weeks later. Both groups will log symptoms daily and receive either UC or SCH-NP care for the 12 week study period.

The UC group will report daily neuropathy symptoms via the web, app or automated phone system and will receive usual care for CIPN symptoms from their existing treatment team. The SCH-NP group will report symptoms similarly but concerning symptoms will trigger a call back from a nurse practitioner who can provide treatment based on standardized algorithmic CIPN guidelines.

In person study visits will take place at baseline and 6 and 12 weeks after randomization. CIPN specific QoL and disability measures, validated CIPN sign scales and detailed information on opioids, neuropathic pain medications and other CIPN treatments will be collected at each visit.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Age ≥ 18.
2. Completion of taxane, platinum, vinca alkaloid-based chemotherapy, bortezomib, thalidomide, lenalidomide, ixazomib, or brentuximab vedotin for cancer in the last 540 days, or ongoing maintenance therapy with bortezomib, thalidomide, lenalidomide or ixazomib for > 90 days.
3. Development of CIPN during or within 3 months of the most recently completed chemotherapy or previous neurotoxic chemotherapy for the same malignancy. For patients on ongoing maintenance therapy: Development of CIPN during current neurotoxic chemotherapy with bortezomib, thalidomide, lenalidomide, ixazomib brentuximab vendotin or vincristine. CIPN diagnosis will be based on clinical diagnosis and the Toronto Criteria for Probable Distal Symmetric Polyneuropathy including the upper and lower extremities.

   The Toronto Criteria for Probable Distal Symmetric Polyneuropathy is defined as a combination of symptoms and signs of neuropathy including:
   1. At least 1 (one) of the following neuropathic symptoms: "asleep numbness", prickling or stabbing, burning or aching pain AND
   2. At least 1 (one) of the following: decreased distal sensation, or unequivocally decreased or absent ankle reflexes. (59)

   Clinical Diagnosis:

   a. Confirmation of CIPN diagnosis by CIPN expert (investigator/co-infestigator based on chart review +/- inperson/virtual interview with examination).
4. Presence of at least one positive neuropathic sensory symptom on the NTSS-6 ranked as moderate or severe on the day of screening or in the preceding week based on recall.
5. The ability to speak/ read sufficient English to be able to communicate with study NP over the phone, utilize the App, website and phone tree (all of which are only available in English).

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Expected treatment with another neurotoxic chemotherapy within the 13 week overall study duration (For example, platinum, taxane, vinca alkaloid, thalidomide, brentuximab vedotin or related drug, or arsenic trioxide. This exclusion does not apply to continuation of treatment for patients on maintenance therapy as described in the inclusion criteria).
2. Presence of a neurological problem that would confound CIPN assessment (lumbar or cervical radiculopathy, or pre-existing neuropathy from another cause such as diabetes).
3. Currently receiving treatment at a pain clinic specifically for CIPN pain.
4. Concurrent participation in a different CIPN or pain treatment trial.
5. For women of childbearing potential: Current pregnancy
6. For women of childbearing potential: Unwillingness to use and acceptable form of birth control for the duration of the study. Acceptable forms of birth control include long acting implantable contraception (ie IUDs, Nexplanon), Oral contraception pills, contraception injections, or strict abstinence if it is part of the subject's current lifestyle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The change in NTSS-6 between the run-in and the 12 week study period. | 12 week study period
  The Neuropathy Total Symptoms Score is a the NTSS- 6, a well validated patient reported neuropathy specific outcome measure. Scores range from 0 to 21.96. Higher scores denote worse outcomes

SECONDARY OUTCOMES:
Change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire. Chemotherapy Induced Peripheral Neuropathy 20 (EORTC- CIPN 20): | baseline, 6 weeks, 12 weeks
  The EORTC CIPN 20 is a 20 item CIPN specific quality of life PRO. Scores range from 20 to 80 with higher scores denoting a worse outcome.
The % of participants taking ≥ 50 morphine milligram equivalents (MME)/ day | baseline, 6 weeks, 12 weeks
  MME/day is the CDC recommended method of measuring and comparing opiate use

CONTACTS AND LOCATIONS:
Overall Officials: Noah A Kolb, MD, Principal Investigator — University of Vermont
Locations (3):
- United States (3):
  - University of Utah, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No